CLINICAL TRIAL: NCT01524094
Title: A Randomised Phase-III Study Comparing Cytoreductive Surgery Plus Intraperitoneal Chemotherapy Versus Modern Systemic Chemotherapy in Colorectal Peritoneal Carcinomatosis.
Brief Title: Cytoreduction and Intraperitoneal Chemotherapy Versus Systemic Chemotherapy in Colorectal Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Wilhelm Graf, M.D., Ph.D., M.D., PhD., Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPS-1
Record Dates: First submitted 2012-01-18; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Peritoneal Carcinomatosis
Keywords: colorectal cancer; cytoreductive surgery; intraperitoneal chemotherapy; systemic chemotherapy; Peritoneal Metastatic Disease From the Colon or Rectum
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: CRS plus postop intraperitoneal chemotherapy. (Experimental): Cytoreductive surgery and postoperative intraperitoneal chemotherapy.
  Interventions: Procedure: Cytoreductive surgery (CRS) plus postoperative intraperitoneal chemotherapy (5-fluorouracil, isovorin)
- Arm B: Systemic chemotherapy alone (Active Comparator): Systemic chemotherapy alone
  Interventions: Drug: Systemic chemotherapy alone (oxaliplatin, 5-fluorouracil, isovorin)

INTERVENTIONS:
Drug: Systemic chemotherapy alone (oxaliplatin, 5-fluorouracil, isovorin) — Oxaliplatin 100 mg/ m2 as a 2 h iv infusion + 5-fluorouracil 400 mg/ m2 iv bolus + Isovorin 100 mg/ m2 as a 2 h infusion followed by 5-fluorouracil 2400 mg/ m2 as a 46 h infusion. Each cycle is given every other week until 12 cycles have been administered.
  Arms: Arm B: Systemic chemotherapy alone
Procedure: Cytoreductive surgery (CRS) plus postoperative intraperitoneal chemotherapy (5-fluorouracil, isovorin) — Cytoreductive surgery has the goal of completely resecting all visible tumor tissue in the abdomen. Sequential postoperative intraperitoneal chemotherapy has the purpose of an adjuvant treatment to eradicate microscopic residual tumor and prevent recurrences in the abdomen. The chemotherapy regimen consisted of intraperitoneal 5-fluorouracil 550 mg/ m2 and intravenous isovorin 30 mg/ m2 day 1-6 med cycles every 4-6 weeks. Six cycles were planned.
  Arms: Arm A: CRS plus postop intraperitoneal chemotherapy.

SUMMARY:
The purpose of this study is to see if there is a difference in survival between two different treatment strategies for colorectal peritoneal surface disease. The control arm administered the currently considered standard treatment which is palliative systemic chemotherapy. The experimental arm received the combination treatment cytoreductive surgery and intraperitoneal chemotherapy. The investigators hypothesis is that the combination treatment will improve the overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease to the peritoneum from colon or rectum (at least two isolated sites of disease)
* verified primary tumor of adenocarcinoma of the colon or rectum
* Potential resectability as judged by the treating surgeon
* Patient is available for follow-up according to the study protocol
* Signed informed consent

Exclusion Criteria:

* Extraabdominal metastases or liver metastases
* Paraaortic or other inoperable lymph node metastases
* Clear indication for surgery only (such as obstruction, bleeding or peritonitis)
* Prior treatment of either arm in the study
* Clinical or histopathological diagnosis of Peritoneal Pseudomyxoma
* Age > 80
* Contraindications for chemotherapy
* Pregnancy or breastfeeding
* Ongoing infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-06; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 8 years

SECONDARY OUTCOMES:
progression free survival | 8 years
Time to secondary treatment | 8 years
Radical resectability | 5 years
Quality of life | 7 years
Health costs | 8 years
Side effects of treatment | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Graf, M.D. Ph.D, Principal Investigator — Uppsala University
Locations (1):
- Akademiska Sjukhuset (Uppsala University Hospital), Uppsala, Sweden

REFERENCES:
- [Background] Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA. Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol. 2003 Oct 15;21(20):3737-43. doi: 10.1200/JCO.2003.04.187. PMID 14551293
- [Background] Assersohn L, Norman A, Cunningham D, Benepal T, Ross PJ, Oates J. Influence of metastatic site as an additional predictor for response and outcome in advanced colorectal carcinoma. Br J Cancer. 1999 Apr;79(11-12):1800-5. doi: 10.1038/sj.bjc.6690287. PMID 10206296
- [Background] Shepherd NA, Baxter KJ, Love SB. The prognostic importance of peritoneal involvement in colonic cancer: a prospective evaluation. Gastroenterology. 1997 Apr;112(4):1096-102. doi: 10.1016/s0016-5085(97)70119-7. PMID 9097991
- [Background] Graf W, Glimelius B, Pahlman L, Bergstrom R. Determinants of prognosis in advanced colorectal cancer. Eur J Cancer. 1991;27(9):1119-23. doi: 10.1016/0277-5379(91)90307-y. PMID 1835620
- [Background] Elias D, Blot F, El Otmany A, Antoun S, Lasser P, Boige V, Rougier P, Ducreux M. Curative treatment of peritoneal carcinomatosis arising from colorectal cancer by complete resection and intraperitoneal chemotherapy. Cancer. 2001 Jul 1;92(1):71-6. doi: 10.1002/1097-0142(20010701)92:13.0.co;2-9. PMID 11443611
- [Background] Saltz LB, Cox JV, Blanke C, Rosen LS, Fehrenbacher L, Moore MJ, Maroun JA, Ackland SP, Locker PK, Pirotta N, Elfring GL, Miller LL. Irinotecan plus fluorouracil and leucovorin for metastatic colorectal cancer. Irinotecan Study Group. N Engl J Med. 2000 Sep 28;343(13):905-14. doi: 10.1056/NEJM200009283431302. PMID 11006366
- [Derived] Cashin PH, Mahteme H, Spang N, Syk I, Frodin JE, Torkzad M, Glimelius B, Graf W. Cytoreductive surgery and intraperitoneal chemotherapy versus systemic chemotherapy for colorectal peritoneal metastases: A randomised trial. Eur J Cancer. 2016 Jan;53:155-62. doi: 10.1016/j.ejca.2015.09.017. Epub 2016 Jan 2. PMID 26751236